CLINICAL TRIAL: NCT05631041
Title: The Possible Anticancer Effect of Silymarin in Patients With Metastatic Colorectal Cancer Receiving Chemotherapy.
Brief Title: Effect of Silymarin in Metastatic Colorectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shimaa Yassin Abdelghafaar Mohamed, principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Silymarin in Colorectal Cancer
Record Dates: First submitted 2022-11-08; First posted 2022-11-30 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Silymarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group I (Control group ; n=32) which will receive FOLFIRI regimen (5-flourouracil, leucovorin, irinotecan) or XELIRI (Capecitabine and irinotecan) with or without target therapy (Bevacizumab).
- Silymarin group (Active Comparator): Group II: (Silymarin group ; n=32) which will receive FOLFIRI regimen (5-flourouracil, leucovorin, irinotecan) or XELIRI (Capecitabine and irinotecan) with or without target therapy (Bevacizumab). plus silymarin 140 mg once daily.
  Interventions: Drug: Silymarin

INTERVENTIONS:
Drug: Silymarin — participants in silymarin group will receive silymarin 140 mg once daily.
  Arms: Silymarin group

SUMMARY:
this work is aim to assess the antitumor effect of silymarin in patients with metastatic colorectal cancer receiving chemotherapy with or without target therapy (Bevacizumab).

DETAILED DESCRIPTION:
Colorectal cancer (CRC) ranks as the third most common cancer globally and second in terms of mortality . Although CRC incidence rates are higher in high-income compared with low-to-middle-income countries (LMICs), mortality is higher in LMICs.

Extensive research within the last decade has shown that silymarin can suppress the proliferation of a variety of tumor cells; this is accomplished through cell cycle arrest at the G1/S-phase, induction of cyclin-dependent kinase inhibitors, down-regulation of anti- apoptotic gene products, inhibition of cell-survival kinases and inhibition of inflammatory transcription factors (e.g., Nuclear Factor- kappa B) through suppression of Nuclear Factor- kappa B-regulated gene products, including Cyclooxygenase-2, Lipoxygenase, Tumor necrosis factor and Interleukin-1. Silymarin can also down-regulate gene products involved in the proliferation of tumor cells (Epidermal Growth Factor Receptor, Cyclooxygenase-2), invasion (Matrix metallopeptidase 9), angiogenesis (Vascular Endothelial growth Factor) and metastasis (adhesion molecules). Silymarin was reported to alter the expression of apoptosis-related proteins including BCL2 associated X protein to induce apoptosis in human gastric cancer cells in a concentration-dependent manner. Silymarin has also been shown to sensitize tumors to chemotherapeutic agents through down-regulation of the Multidrug resistance protein and other mechanisms. In addition to its chemo-preventive effects, silymarin exhibits antitumor activity against human tumors in rodents. so we aim to assess the antitumor activity of silymarin in metastatic colorectal cancer patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with histologically and/or radiologically confirmed diagnosis of metastatic colorectal carcinoma.
* Patients who received FOLFOX or XELOX as first line chemotherapy
* Both genders.
* Age ≥18 years old.
* Performance status 0-1 according to the Eastern Cooperative Oncology Group (ECOG).
* Patients with adequate hematologic parameters (white blood cell count

  ≥3000/mm3, granulocytes ≥1500/mm3, platelets ≥100,000/mm3, hemoglobin ≥ 8 gm/l).
* Patients with adequate renal functions (serum creatinine ≤1.5 mg/dL).
* Patients with adequate hepatic functions (bilirubin ≤1.5 mg/dL or albumin ≥3 g/dL).

Exclusion Criteria:

* - Patients with active liver diseases (chronic viral hepatitis, autoimmune hepatitis, alcoholic hepatitis, Wilson's disease, hemochromatosis, or cirrhosis).
* Patients with a history of other malignancy.
* Patients with brain metastasis.
* Patients with active infection.
* Patients with RAS wild type cancer.
* Patients on chronic use of corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The change between groups in response rate (RECIST) | At baseline, pre-intervention and at the end of last chemotherapy cycle ( 3 months from the beginning ) patients will recieve either Folfiri 6 cycles ( each cycle is 14 days) or Xeliri 4 cycles ( each cycle is 21 days)
  Tumor response is characterized by both objective response rates (ORR=Complete response + partial response) and disease control rate (DCR= complete response + partial response + stable disease). In addition, complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) will be evaluated.
  Follow-up for one year will be carried out to determine progression free survival (PFS) and the overall survival (OS) or one year survival.

SECONDARY OUTCOMES:
Changes in serum levels of the measured biological marker serum carcinoembryonic antigen in ng/ ml or Carbohydrate antigen 19-9 in U/ml. | 3 Months. At baseline( pre-intervention )and at the end of last chemotherapy cycle ( 3 months from the beginning ) patients will recieve either Folfiri 6 cycles ( each cycle is 14 days) or Xeliri 4 cycles ( each cycle is 21 days).
  As Tumor Marker if the baseline is elevated.
Changes in serum levels of the measured biological marker serum vascular endothelial growth factor in pg/ml. | 3 Months. At baseline( pre-intervention )and at the end of last chemotherapy cycle ( 3 months from the beginning ) patients will recieve either Folfiri 6 cycles ( each cycle is 14 days) or Xeliri 4 cycles ( each cycle is 21 days).
  As a marker of angiogenesis.
Changes in serum levels of the measured biological marker serum Bax protein in ng/ml. | 3 Months. At baseline( pre-intervention )and at the end of last chemotherapy cycle ( 3 months from the beginning ) patients will recieve either Folfiri 6 cycles ( each cycle is 14 days) or Xeliri 4 cycles ( each cycle is 21 days).
  As a marker for apoptosis.
Changes in serum levels of the measured biological marker serum permeability glycoprotein in ng/ml | 3 Months. At baseline( pre-intervention )and at the end of last chemotherapy cycle ( 3 months from the beginning ) patients will recieve either Folfiri 6 cycles ( each cycle is 14 days) or Xeliri 4 cycles ( each cycle is 21 days).
  As a marker for chemo-sensitization.

CONTACTS AND LOCATIONS:
Overall Officials: shimaa yassin, pharmacist, Principal Investigator — Tanta University; Tarek Mostafa, professor, Study Director — Tanta University; Sahar Elhaggar, professor, Study Director — Tanta University; Mohammed Alam El-Din, professor, Study Director — Tanta University
Locations (1):
- faculty of Pharmacy , Tanta University, Tanta, Egypt

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Abou-Zeid AA, Khafagy W, Marzouk DM, Alaa A, Mostafa I, Ela MA. Colorectal cancer in Egypt. Dis Colon Rectum. 2002 Sep;45(9):1255-60. doi: 10.1007/s10350-004-6401-z. PMID 12352245
- [Background] Agarwal R, Agarwal C, Ichikawa H, Singh RP, Aggarwal BB. Anticancer potential of silymarin: from bench to bed side. Anticancer Res. 2006 Nov-Dec;26(6B):4457-98. PMID 17201169
- [Background] Kim SH, Choo GS, Yoo ES, Woo JS, Han SH, Lee JH, Jung JY. Silymarin induces inhibition of growth and apoptosis through modulation of the MAPK signaling pathway in AGS human gastric cancer cells. Oncol Rep. 2019 Nov;42(5):1904-1914. doi: 10.3892/or.2019.7295. Epub 2019 Aug 28. PMID 31485597
- [Background] Alcaide J, Funez R, Rueda A, Perez-Ruiz E, Pereda T, Rodrigo I, Covenas R, Munoz M, Redondo M. The role and prognostic value of apoptosis in colorectal carcinoma. BMC Clin Pathol. 2013 Oct 10;13(1):24. doi: 10.1186/1472-6890-13-24. PMID 24106912